CLINICAL TRIAL: NCT02215759
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 44370 TA Tablets (100 mg, 200 mg and 300 mg Three Times Every Two Hours on One Day and q.d. for Another 2 to 3 Days) in Healthy Male and Female Volunteers, a Randomised, Doubleblind, Placebo-controlled Within Dose Groups Phase I Study
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 44370 TA Tablets in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1246.15
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 44370 TA (Experimental)
  Interventions: Drug: BI 44370 TA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 44370 TA
  Arms: BI 44370 TA
Drug: Placebo
  Arms: Placebo

SUMMARY:
Evaluation of safety, tolerability and pharmacokinetics of multiple rising oral doses of BI 44370 TA in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria based upon a complete medical history, including the physical examination, vital signs, 12-lead ECG, clinical laboratory tests
* Age ≥21 and Age ≤50 year
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including vital signs and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoking (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

Exclusion criteria for male subjects are:

* Not willing to use adequate contraception (condom plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

Exclusion criteria for female subjects are:

* Pregnancy or planning to become pregnant within 3 months of study completion
* Positive pregnancy test
* No adequate contraception, e.g. implants, injectables, combined oral contraceptives, surgical sterilisation (including hysterectomy or bilateral ovariectomy), intrauterine device, not having used an adequate method of contraception for at least three months prior to participation in the study, and not willing or able to use such adequate contraception until three months after the last intake of study drug
* Lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 36 days
Number of patients with clinically relevant findings in vital signs | up to 7 days after last drug administration
Number of patients with clinically relevant findings in 12-lead ECG (electrocardiogram) | up to 7 days after last drug administration
Number of patients with clinically relevant laboratory findings | up to 7 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 7 days after last drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax ) for several time points | up to 4 days
Time from dosing to maximum measured concentration of the analyte in plasma (tmax) for several time points | up to 4 days
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC) for several time points | up to 4 days
The percentage of the AUC 0-∞ that is obtained by extrapolation (%AUCtz-∞) for several time points | up to 4 days
Terminal rate constant in plasma (λz) for several time points | up to 4 days
Terminal half-life of the analyte in plasma (t1/2) for several time points | up to 4 days
Mean residence time of the analyte in the body after p.o. administration (MRTpo) for several time points | up to 4 days
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) for several time points | up to 4 days
Apparent volume of distribution during the terminal phase λz following an extravascular administration (Vz/F) for several time points | up to 4 days
Amount of analyte that is eliminated in urine from zero to 24 h after drug administration (Ae0-24) for several time points | up to 4 days
Fraction of analyte eliminated in urine from zero to 24 h after drug administration (fe0-24) for several time points | up to 4 days
Renal clearance of the analyte from zero to 24 h after drug administration (CLR,0-24) for several time points | up to 4 days
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 4 days
Accumulation ratio (RA) based on Cmax for several time points | up to 4 days
RA based on AUC for several time points | up to 4 days
Linearity index (LI) of the analyte in plasma | up to 4 days